CLINICAL TRIAL: NCT04536532
Title: A Single-center, Randomized, Double-blind, Single and Multiple Dosing, Evaluation HEC121120 Tolerance in Healthy Subjects and Patients With Chronic Hepatitis B, Pharmacokinetics Characteristics and Antiviral Activity of Ⅰ Phase of Study
Brief Title: Evaluation HEC121120 Tolerance in Healthy Subjects and Patients With Chronic Hepatitis B, Pharmacokinetics Characteristics and Antiviral Activity of Ⅰ Phase of Study
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company decision to discontinue trial
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC121120-P-01
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HEC121120 tablets (Experimental): part 1(Health volunteer): single-Dose Study: There will be a total of 6 dose cohorts: 25 mg、50 mg、100 mg、400 mg、600 mg、800 mg food effect：200 mg multiple-dose study: 200 mg part 2(Patients with chronic hepatitis B): There will be a total of 3 dose cohorts:100、200、400 mg
  Interventions: Drug: HEC121120 tablets
- HEC121120 placebo tablets (Placebo Comparator): part 1(Health volunteer): single-Dose Study: There will be a total of 6 dose cohorts: 25 mg、50 mg、100 mg、400 mg、600 mg、800 mg food effect：200 mg multiple-dose study: 200 mg part 2(Patients with chronic hepatitis B): There will be a total of 3 dose cohorts:100、200、400 mg
  Interventions: Drug: HEC121120 placebo tablets
- entecavir tablets (Active Comparator): part 2(Patients with chronic hepatitis B): 0.5 mg
  Interventions: Drug: entecavir tablets
- entecavir placebo tablets (Placebo Comparator): part 2(Patients with chronic hepatitis B): 0.5 mg
  Interventions: Drug: entecavir placebo tablets

INTERVENTIONS:
Drug: HEC121120 tablets — single-Dose Study: Each dose of HEC121120 and placebo will be administered with approximately 240 mL of water in the morning after fasting for at least 10 hours overnight.
  multiple-dose study/Patients with chronic hepatitis B:The study doses, administration method (fasted or fed), dosing frequency, and dosing period are all to be determined based on data from the single-dose study and/or multiple-dose study.
  Arms: HEC121120 tablets
Drug: HEC121120 placebo tablets — single-Dose Study: Each dose of HEC121120 and placebo will be administered with approximately 240 mL of water in the morning after fasting for at least 10 hours overnight.
  multiple-dose study/Patients with chronic hepatitis B:The study doses, administration method (fasted or fed), dosing frequency, and dosing period are all to be determined based on data from the single-dose study and/or multiple-dose study.
  Arms: HEC121120 placebo tablets
Drug: entecavir tablets — Patients with chronic hepatitis B：Administered Entecavir orally once daily for consecutive 28 days in fasted state
  Arms: entecavir tablets
Drug: entecavir placebo tablets — Patients with chronic hepatitis B：Administered Entecavir placebo orally once daily for consecutive 28 days in fasted state
  Arms: entecavir placebo tablets

SUMMARY:
The Safety, Tolerability, Pharmacokinetics and antiviral activity Study of Anti hepatitis B virus treatment drug HEC121120 in Healthy subjects and in patients with chronic hepatitis B

DETAILED DESCRIPTION:
This study consists of two parts: healthy subjects and chronic hepatitis B patients. Healthy subjects will conduct a single-dose, multiple-dose and food effect study.

I. Single-Dose Study：There will be a total of 6 dose cohorts（25 mg, 50 mg, 100 mg, 400 mg, 600 mg, 800 mg). 25 mg cohort as experimental cohort, plans to enroll 4 subjects (male or female) who will use HEC121120 tablets . The other else cohorts will include 10 subjects, of which 8 receives HEC121120 tablets and 2 receives placebo, regardless of gender. Each subject will only participate in one dose cohort. Each cohort will be divided into 2 group. The first group consists of 3 sentinels, two receiving active and one placebo. The second group will consist of the remainder of the cohort (6 active and 1 placebo) and, following review of the available safety data, will be dosed 24 hours after the sentinel group. Subjects can leave the pharmacy after their biological samples are collected on day 5. Subjects in each cohort will receive a single dose of HEC121120 or placebo in the fasted state on day 1, and safety evaluation is to be performed on day 2 and 5.

II. Food effect: There will be 1 dose cohort (200 mg), only to be admitted to the 100 mg dose cohort if a single dose has been completed and is safe and well tolerated. A total of 18 subjects were enrolled in this dose cohort, divided into two groups A and B (9 subjects in each group, 8 subjects in each group received HEC121120 and 1 received the placebo, with the ratio of male to female as close as possible. All subjects were required to participate in a single dose and food influence study on pharmacokinetics. Two cycles of cross-dose administration were performed, with a washout period of 7 days. Four sentinels were first enrolled in group A, and their safety indexes were evaluated by the investigator at least 24 h after administration. If tolerated, the remaining 5 sentinels could be enrolled in group A, and the remaining 4 sentinels could be enrolled in group B. The safety indexes were evaluated by the investigator at least 24 h after administration, if tolerated, the remaining 5 sentinels could be enrolled in group B.

III. Multi-Dose Study: There will be 1 dose(200 mg) cohort which will consist of 12 subjects, of which 10 receive HEC121120 tablets and 2 receive placebo, with the ratio of male to female as close as possible. All subjects will receive HEC121120 or placebo for 5 consecutive days (study doses, administration method (fasted or fed), dosing frequency, and dosing period are all to be determined based on data from the single-dose study and multiple-dose study). Subjects can leave pharmacy after their biological samples are collected. Safety evaluation is to be performed on day 3 and 7.

IV:Chronic hepatitis B patients: There will be a total of 3 dose cohorts (100、200、400 mg). Each cohort will consist of 14 subjects, of which 12 receive HEC121120 tablets and placebo(Entecavir simulation tablet), 2 receive Entecavir and placebo(HEC121120 simulation tablet). It is necessary to determine the administration method and dose for patients with chronic hepatitis B based on the results of the tolerance and PK study of healthy subjects. Each subject will only participate in one dose cohort.Initially, the drug frequency was set as once a day for 28 consecutive days. Safety and antiviral activity evaluation is to be performed on day 7, 14, 21±2, 29, 35±2.

ELIGIBILITY:
Health volunteer

Inclusion Criteria:

1. Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions.
2. Be able to complete the study according to the trail protocol.
3. Subjects (including partners) have no pregnancy plan within 6 months after the last dose of study drug and voluntarily take effective contraceptive measures.
4. subjects and must be 18 to 45 years of age inclusive.
5. Body weight ≥ 45 kg and body mass index（BMI）between 18 and 28 kg / m^2, inclusive.
6. Physical examination and vital signs without clinically significant abnormalities.

Exclusion Criteria:

1. Use of >5 cigarettes per day during the past 3 months.
2. Known history of allergy to study drugs，or allergies constitution ( multiple drug and food allergies).
3. History of alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits or 100 mL of wine).
4. Donation or loss of blood over 450 mL within 3 months prior to screening. 5.12-lead ECG with clinically significant.

6.Positive for Viral hepatitis (including hepatitis B and C), HIV and syphilis. 7.Subjects deemed unsuitable by the investigator for any other reason.

Patients with chronic hepatitis B

Inclusion Criteria:

1. Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions.
2. Be able to complete the study according to the trail protocol.
3. Subjects (including partners) have no pregnancy plan within 6 months after the last dose of study drug and voluntarily take effective contraceptive measures.
4. subjects and must be 18 to 65 years of age inclusive.
5. Body mass index（BMI）between 18 and 32 kg / m^2, inclusive.
6. There is evidence of hepatitis B infection for more than 6 months。
7. HBV DNA copies≥2.0×10^4 IU/mL.
8. ALT≤5×ULN，TBIL≤2×ULN
9. No cirrhosis.

Exclusion Criteria:

1. Use of >5 cigarettes per day during the past 3 months.
2. Known history of allergy to study drugs，or allergies constitution ( multiple drug and food allergies).
3. Female subjects were lactating or had positive serum pregnancy results during the screening or testing period.
4. Donation or loss of blood over 450 mL within 3 months prior to screening. 5.12-lead ECG with clinically significant.

6.Positive for Viral hepatitis C, HIV and syphilis. 7. AFP>50 ng/mL. 8. eGFR<60 mL/min/1.73m^2 9.Subjects deemed unsuitable by the investigator for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-03-12 (Actual); Study Completion 2023-03-12 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Time Frame: From Days 1-35
  Incidence of adverse events
Cmax | Time Frame: Day 1-7
  Maximum plasma concentration of study drugs
AUC | Time Frame: Day 1-7
  Maximum plasma concentration of study drugs
HBV DNA | Time Frame: Day 29-35
  Hepatitis B virus DNA

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Jilin, Changchun, China